CLINICAL TRIAL: NCT05658744
Title: Effect Of Reducing Insulin Implementation Errors In Education Compared To Routine Approach In Type 2 Diabetes Patients Using Insulin: A Randomized Controlled Study
Brief Title: Video Training to Reduce Insulin Administration Errors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Principal Investigator, Gunes Feyizoglu, Principal Investigator, Goztepe Prof Dr Suleyman Yalcın City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SuleymanYalcın
Record Dates: First submitted 2022-12-03; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Injection Pad; Injection Site; Insulin Implementation Errors; Educational Problems
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Masking Description: Blinding of patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video group (Experimental): Insulin administration video was shown to 52 patients with diabetes using insulin. The video was sent to the patients' mobile phones
  Interventions: Behavioral: Video group
- Brochure group (Experimental): Insulin administration leaflet was given to 42 patients with diabetes using insulin. Patients read the brochure aloud
  Interventions: Behavioral: Video group

INTERVENTIONS:
Behavioral: Video group — Insulin administration video was sent to the mobile phones of the patients assigned to the video group

SUMMARY:
Efficiency of training with video to reduce injection errors in patients using insulin

DETAILED DESCRIPTION:
The aim of this study is to examine the effects of using insulin administration video and insulin administration brochure as teaching materials in insulin administration training given to type 2 diabetes patients on correcting insulin administration errors. This randomized controlled experimental study was carried out with 94 people who applied to the diabetes outpatient clinic of Istanbul Medeniyet University Goztepe Training and Research Hospital between December 2019 and January 2021. Using a computer-based randomization method, 52 and 42 people were assigned to the groups that received training with video and brochures, respectively. In the first interview, patients' insulin administration characteristics were evaluated, and the training was repeated using the video or brochure, after which the training material corresponding to the group according to the randomization list was given. Insulin administration characteristics of the patients were re-evaluated one week and three months later. Patient information form developed by the researcher based on the literature was used to collect the data. Data were analysed using descriptive statistics, independent sample t-test and Mann Whitney U test. The error rates in the interviews were analysed with the Cochrane Q test, and the relationship between independent categorical variables was examined with the Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* mobile phone can download video
* video watching skills

Exclusion Criteria:

* illiterate patient
* new to insulin therapy
* who can't watch video on mobile phone

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-12-25 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Behavior change | 3 months later
  Video training is effective in reducing insulin administration errors. There was no statistically significant difference between the groups in terms of sociodemographic characteristics of the individuals in the video and brochure group (p>0.05). The mean number of corrects in insulin administration increased from 12.94 to 20.15 in the group given the training video and from 14.33 to 18.67 in the group given the training brochure, with the patients who received video training having a higher mean number of corrects than the patients who received training with a brochure (t=2.69, p=0.009). In conclusion, retraining patients using insulin therapy with a video was found to be an effective approach to reduce insulin administration errors.

CONTACTS AND LOCATIONS:
Locations (1):
- Goztepe Prof Dr Suleyman Yalcın City Hospital, Kadıköy, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Feyizoglu GA, Can G. Injection Errors Are Still Common in Insulin Therapy! Could It be a Solution? J Eval Clin Pract. 2025 Jun;31(4):e70156. doi: 10.1111/jep.70156. PMID 40545932